CLINICAL TRIAL: NCT04320628
Title: Randomized Double-Blind Controlled Clinical Trial Comparing Sodium Hypochlorite Antiseptic to Normal Saline in Reducing Bioburden in Wounds
Brief Title: Randomized Double-Blind Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Anacapa Technologies Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANTISEPTIC1
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Chronic Wounds; Acute Wounds

STUDY DESIGN:
Intervention Model Description: AnaSept® AnaSept® Antimicrobial Skin and Wound Cleanser is a clear liquid consisting of 0.057% sodium hypochlorite (NaOCl) in an isotonic saline.
Who Masked: Participant, Investigator
Masking Description: This protocol is double-blinded. Subjects will be randomized 1:1 to have their wound cleansed with either NSS or NaOCl. Unblinded staff will prepare the solutions for the two arms the morning of the day of enrollment. NSS and NaOCl will be placed in labeled containers consistent with the randomization scheme. NaOCl has a faint odor of chlorine. In order to maintain the blind the containers will have chlorine placed on the outside of bottom of the container and in the treatment room an open container of chlorine bleach will be safely positioned as to avoid injury to subjects and research personnel, but close enough to provide a mild chlorine smell in the room. Finally, the unblinded research staff will provide the subject with their 4-week supply of NSS or NaOCl to take home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental (Experimental): Target ulcer cleansed with NaOCl. After cleansing the wound a second MiX is performed. The subject is given a four-week supply of NaOCl.
  Interventions: Device: AnaSept®
- Control (Placebo Comparator): Target ulcer cleansed with NSS. After cleansing the wound a second MiX is performed. The subject is given a four-week supply of NSS.
  Interventions: Other: NSS

INTERVENTIONS:
Device: AnaSept® — AnaSept® AnaSept® Antimicrobial Skin and Wound Cleanser is a clear liquid consisting of 0.057% sodium hypochlorite (NaOCl) in an isotonic saline. It has a broad-spectrum of antimicrobial action inhibiting the growth of Staphlyococcus aureus, Psuedomonas aeruginosa, Escherichia coli, Proteus mirabilis, Serratia marcescens, Clostridium difficile, including antibiotic resistant Methicillin Resistant Staphylococcus aureus (MRSA), Vancomycin Resistant Enterococcus faecalis (VRE), Carbapenem Resistant E.coli (CRE) and Acinetobacter baumannii, that are commonly found in wound bed as well as fungi such as Candida albicans and Aspergillus niger. However, NaOCL is non-toxic to mammalian cells.
  Other Names: ANTISEPTIC
  Arms: Experimental
Other: NSS — NSS
  Arms: Control

SUMMARY:
The study is a randomized double-blind controlled clinical trial designed to compare the ability of NaOCl to NSS in the reduction of bacterial burden in nonhealing acute and chronic wounds.

DETAILED DESCRIPTION:
The study is a randomized double-blind controlled clinical trial designed to compare the ability of NaOCl to NSS in the reduction of bacterial burden in nonhealing acute and chronic wounds. Using the generally accepted surrogate endpoint of surface area reduction at 4 weeks, the study will also compare the healing of subjects utilizing NaOCl vs. NSS.

After consenting, the ulcers of eligible subjects are measured, photographed and undergo the MolecuLight imaging procedure (MiX). The subject is then randomized to one of two arms: target ulcer cleansed with NaOCl or NSS. After cleansing the wound a second MiX is performed. The subject is given a four-week supply of either NaOCl or NSS.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with acute or chronic wounds that have been present for a minimum of 4 weeks.
2. A signed and dated informed consent form.
3. Subject is willing and able to comply with instructions and scheduled visits.

Exclusion Criteria:

1. The Subject has other concurrent conditions that in the opinion of the Investigator may compromise subject safety.
2. The subject's wound has not been present for at least 4 weeks.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Reduction in bacterial bioburden | 4 weeks
  The reduction in bacterial bioburden as determined by the MolecuLight Procedure (MiX) between normal saline (NSS) and sodium hypochlorite (NaOCl) wound washing.

SECONDARY OUTCOMES:
Healing rate | 4 weeks
  The effect on healing (surface area reduction) at a surrogate endpoint of 4 weeks between wounds washed with NaOCl vs wounds washed with NSS.
Pain Score (PEG) | 4 weeks
  PEG Scale Assessing Pain Intensity and Interference (Pain, Enjoyment, General Activity) The difference in pain scores (PEG) between subjects treated with NaOCl vs, NSS.It consists of three 1-10 rating scales: numerical, enjoyment of life and general activity.
  The subject indicates a numerical value that best represents the pain intensity at ulcer site on a scale of 0 to 10 anchored by word descriptors at each end, as "no pain" on the left side and "Pain as bad as you can imagine" on the right side of the number line. The number 0 represents "no pain", the number 5 represents "moderate pain" and the number 10 represents the "worst possible pain".
Adverse Events | 4 weeks
  The difference in adverse events between subjects treated with NaOCl vs, NSS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD,FACS, Principal Investigator — Serena Group
Locations (1):
- Serena Group Research Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share